CLINICAL TRIAL: NCT05769738
Title: The Addition of Inhaled FUROsemide to Standard of Care in COPD Exacerbation: a Randomized Double Blinded Control Trial (FUROSCOPE Trial)
Brief Title: The Addition of Inhaled Furosemide to Standard Treatment of COPD Exacerbation
Acronym: FUROSCOPE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2022-0187
Record Dates: First submitted 2023-02-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation; COPD Exacerbation
Keywords: COPD; furosemide; dyspnea; inhaled furosemide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Furosemide; Diuretics; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both medications will be prepared by the pharmacists, the only unblinded personnel in the study, as transparent solutions in similar syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide group (Experimental): Inhaled furosemide
  Interventions: Drug: Furosemide
- Placebo group (Placebo Comparator): Inhaled saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Furosemide — 40mg (4ml) of furosemide to be nebulized 3 times daily for 3 days
  Other Names: Lasix; Diuretic
  Arms: Furosemide group
Drug: Normal saline — 4ml of normal saline to be nebulized 3 times daily for 3 days
  Arms: Placebo group

SUMMARY:
The goal of this randomized controlled trial is to determine the effect of adding inhaled furosemide to the known treatment of patient with Chronic obstructive pulmonary disease (COPD) exacerbation. It primarily aims at studying its effect on:

1. Relief of dyspnea sensation
2. Length of hospital stay

Participants will be receiving the standard therapy of COPD exacerbation plus either inhaled furosemide or inhaled saline over 3 days. They will be asked to:

* Perform spirometry
* Fill in dyspnea score
* Do arterial blood gases (ABGs)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with COPD
* Presenting with COPD exacerbation
* Requiring hospitalization

Exclusion Criteria:

* Hemodynamically instability (systolic blood pressure ≤ 90mmHg, heart rate ≥ 120 or ≤ 50 Bpm)
* Decreased level of consciousness
* Non-invasive mechanical ventilation or intubation at the time of recruitment
* >5 liters of oxygen at the time of recruitment
* Pregnant patients
* Other primary pulmonary disease or heart failure exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in dyspnea score from baseline as assessed by visual analogue scale (VAS) | at 24 hours
  Visual analogue scale is a scale from 0 to 10, where 0 means no dyspnea at all and 10 is the worse dyspnea ever
Change in dyspnea score from baseline as assessed by visual analogue scale (VAS) | at 72 hours
  Visual analogue scale is a scale from 0 to 10, where 0 means no dyspnea at all and 10 is the worse dyspnea ever
Change in length of hospital stay | From admission to hospital discharge, up to 1 year

SECONDARY OUTCOMES:
Change in lung volumes from baseline as measured by bedside spirometer | On days 0, 1 and 3
  Forced expiratory volume in first second (FEV1) and forced vital capacity (FVC)
Change in Arterial blood gases | On days 0 and 1
Change in heart rate from baseline | On days 0, 1 and 3
Change in systolic and diastolic blood pressure from baseline | On days 0, 1 and 3
Change in steroid dose | Through hospital stay, up till 1 year
Change in the number of patients requiring intubation or non-invasive mechanical ventilation | Through hospital stay, up till 1 year
  Measured by questionnaire
Change in mortality | Through hospital stay, up till 1 year
Number of patients with adverse events as documented by questionnaires | On days 1,2,3
  Including: kidney injury measured by Creatinine and urine output, electrolyte disturbances (sodium and potassium levels)

CONTACTS AND LOCATIONS:
Overall Officials: Nivine Abou Dargham, MD, Study Director — AUBMC; Salah Zeineddine, MD, Principal Investigator — AUBMC; Hisham Bou Fakhreddine, MD, Principal Investigator — AUBMC

IPD SHARING:
Plan to Share IPD: No